CLINICAL TRIAL: NCT01330368
Title: Spine Quantitative Computed Tomography (QCT) for the Assessment of Osteoporosis on Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 10-007747
Record Dates: First submitted 2010-12-14; First posted 2011-04-06 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; SLE; Lupus; children with SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare healthy children to children who have systemic lupus erythematosus (SLE). SLE is a childhood disease that has high risk for low bone mass and vertebral compression fractures.

DETAILED DESCRIPTION:
The purpose of this research study is to measure bone mass in children with SLE using different measurement techniques. Children with chronic illnesses are at risk of bone fragility. This is important because bone fragility can result in childhood fractures especially children with SLE. Therefore better diagnosis technique can lead to better management of bone health.

ELIGIBILITY:
Inclusion Criteria:

* For SLE subjects: Subjects age 5-21 drawn from rheumatology clinic at Children's Hospital of Philadelphia diagnosed with SLE for at least 1 month. Also subjects with no known vertebral compression fracture of L2.
* For Control subjects: Subjects age 5-21. Controls will be a 50% male/female.

Exclusion Criteria:

* For SLE subjects: Subjects with SLE will be excluded if they have conditions or drug exposure unrelated to SLE and known to impact growth or bone health.
* For Control subjects: Chronic disease or syndrome known to affect growth or bone health, prematurity (<37 weeks gestation), or use of any medication known to affect growth.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 200 control patients (124 controls participated in unique protocol ID: 2007-10-5528 data will be used for this study, we will be trying to recruit about 76 control patients for this study) and 30 study patients with SLE
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Age and sex specific z-scores for lumbar spine (L2) volumetric bone mineral density (BMD) (trabecular and total) and vertebral volume. | 2 years

SECONDARY OUTCOMES:
Mean lumbar spine stiffness and strength in children with SLE and healthy controls correlation between standard and low dose lumbar spine. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jon Burnham, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States